CLINICAL TRIAL: NCT01133314
Title: The Routine Use of Coartem for Treatment of Symptomatic Children With Plasmodium Falciparum in Bissau - 2
Brief Title: Artemether-Lumefantrine Effectiveness in Guinea-Bissau 2
Status: Completed | Type: Observational
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Other Study IDs: AL-eff 2010-2
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2015-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — App 50 - 100 microliters blood on filterpaper for identification of parasite. Furthermore, whenever the health staff use a RDT this will be saved for the same analyses.
Oversight: Data Monitoring Committee: No

SUMMARY:
The routine treatment of children with antimalarials will be monitored. Children with a positive malaria film and/or a positive rapid diagnostic test (RDT) will have a capillary blood sample taken to verify the diagnosis and to monitor the pattern of resistance.

DETAILED DESCRIPTION:
Children from Bissau seeking medical advice and who are recommended treatment for malaria in accordance with the current routines will be included as follows:

All children getting the clinical diagnosis of malaria will be registered and basic information collected.

All children with a positive malaria film and/or a positive RDT will be asked for a capillary blood sample (app. 50 - 100 microliters on a filterpaper). Using PCR the parasitological diagnosis will be verified and if parasites are identified the resistance patterns will be examined. Both the capillary blood samples and the RDTs (if taken by the health staff) will be used in order to examine whether the RDTs can be used for routine monitoring of resistance in an area.

The study does not interfere in the routine treatment of the health staff. None of the children will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Children seeking a health centre and by the health staff given the diagnosis: malaria and/or being treated with an antimalarial.

Exclusion Criteria:

* Children where the parents do not accept to participate in the study.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children seeking a health centre and by the health staff given the diagnosis: malaria and/or being treated with an antimalarial.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of children treated for malaria with a parasitological confirmed malaria. | 6 weeks
  The blood samples will be analysed for parasites at the end of the study. The results do not have any impact on the treatment of the children.

SECONDARY OUTCOMES:
Percentage of the parasites with mutations coding for resistance to antimalarials. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Poul-Erik Kofoed, MD, Ph.d., Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Bissau Codex, Guinea-Bissau